CLINICAL TRIAL: NCT00904839
Title: A Phase I-II Study of BIBF 1120 and FOLFOX Compared to Bevacizumab and FOLFOX in First Line Metastatic Colorectal Cancer Patients
Brief Title: BIBF 1120 Versus Bevacizumab in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.51; 2008-005364-14 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nintedanib; Bevacizumab

ARMS (2):
- BIBF 1120 + mFolfox6 (Experimental): BIBF1120 medium dose twice daily
  Interventions: Drug: BIBF 1120; Drug: mFolfox 6; Drug: bevacizumab
- Bevacizumab + mFolfox6 (Active Comparator): Bevacizumab 5mg/kg once daily every other week
  Interventions: Drug: BIBF 1120; Drug: mFolfox; Drug: Bevacizumab

INTERVENTIONS:
Drug: BIBF 1120 — BIBF 1120 100 and 150 mg capsules
  Arms: BIBF 1120 + mFolfox6
Drug: BIBF 1120 — BIBF 1120 100 and 150 mg capsules
  Arms: Bevacizumab + mFolfox6
Drug: mFolfox — standard i.v chemotherapy
  Arms: Bevacizumab + mFolfox6
Drug: Bevacizumab — 100 mg/Kg solution , IV infusion
  Arms: Bevacizumab + mFolfox6
Drug: mFolfox 6 — IV standard chemotherapy
  Arms: BIBF 1120 + mFolfox6
Drug: bevacizumab — 100 mg/4 ml solution
  Arms: BIBF 1120 + mFolfox6

SUMMARY:
The primary objective of this study is to evaluate PFS rate at 9 months of BIBF 1120 in combination with mFolfox6 compared with mFolfox6 combined to bevacizumab in first line patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion criteria:

1. Age >= 18 years
2. Histologically proven colorectal adenocarcinoma
3. No previous oxaliplatin based chemotherapy is allowed unless disease free survival after the end of chemotherapy > = 12 months
4. No previous therapy with VEGFR or EGFR inhibitors
5. No prior systemic therapy for metastatic CRC
6. No previous adjuvant therapy with fluoropyrimidines is allowed unless disease free survival after the end of chemotherapy > 6 months
7. ECOG performance status < = 2
8. Adequate hepatic, renal and bone marrow functions:
9. No uncontrolled hypertension
10. Signed and dated written informed consent prior to admission to the study

Exclusion criteria:

1. Treatment with any investigational drug within 28 days of trial onset.
2. History of other malignancies in the last 5 years, in particular those that could affect compliance with the protocol or interpretation of results.
3. Serious concomitant disease, especially those affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug,
4. Major injuries and/or surgery or bone fracture within 4 weeks of trial inclusion, or planned surgical procedures during the trial period.
5. Significant cardiovascular diseases
6. History of severe haemorrhagic or thromboembolic event in the past 12 months. Known inherited predisposition to bleeding or to thrombosis.
7. Patient with brain metastases that are symptomatic and/or require therapy.
8. Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (47):
- Belgium (4):
  - 1199.51.32002 Boehringer Ingelheim Investigational Site, Bonheiden
  - 1199.51.32005 Boehringer Ingelheim Investigational Site, Brussels
  - 1199.51.32006 Boehringer Ingelheim Investigational Site, Brussels
  - 1199.51.32001 Boehringer Ingelheim Investigational Site, Leuven
- France (26):
  - 1199.51.3306A Boehringer Ingelheim Investigational Site, Nice
  - 1199.51.3306B Boehringer Ingelheim Investigational Site, Nice
  - 1199.51.3306C Boehringer Ingelheim Investigational Site, Nice
  - 1199.51.3306D Boehringer Ingelheim Investigational Site, Nice
  - 1199.51.3301A Boehringer Ingelheim Investigational Site, Paris
  - 1199.51.3301B Boehringer Ingelheim Investigational Site, Paris
  - 1199.51.3301C Boehringer Ingelheim Investigational Site, Paris
  - 1199.51.3301D Boehringer Ingelheim Investigational Site, Paris
  - 1199.51.3307A Boehringer Ingelheim Investigational Site, Reims
  - 1199.51.3307B Boehringer Ingelheim Investigational Site, Reims
  - 1199.51.3307C Boehringer Ingelheim Investigational Site, Reims
  - 1199.51.3308A Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1199.51.3308B Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1199.51.3308C Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1199.51.3308D Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1199.51.3308E Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 1199.51.3305A Boehringer Ingelheim Investigational Site, Toulouse
  - 1199.51.3305B Boehringer Ingelheim Investigational Site, Toulouse
  - 1199.51.3305C Boehringer Ingelheim Investigational Site, Toulouse
  - 1199.51.3305D Boehringer Ingelheim Investigational Site, Toulouse
  - 1199.51.3305E Boehringer Ingelheim Investigational Site, Toulouse
  - 1199.51.3302A Boehringer Ingelheim Investigational Site, Villejuif
  - 1199.51.3302B Boehringer Ingelheim Investigational Site, Villejuif
  - 1199.51.3302C Boehringer Ingelheim Investigational Site, Villejuif
  - 1199.51.3302D Boehringer Ingelheim Investigational Site, Villejuif
  - 1199.51.3302E Boehringer Ingelheim Investigational Site, Villejuif
- Germany (6):
  - 1199.51.49001 Boehringer Ingelheim Investigational Site, Celle
  - 1199.51.49002 Boehringer Ingelheim Investigational Site, Dresden
  - 1199.51.49003 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1199.51.49004 Boehringer Ingelheim Investigational Site, Halle
  - 1199.51.49006 Boehringer Ingelheim Investigational Site, Mainz
  - 1199.51.49008 Boehringer Ingelheim Investigational Site, Schwäbisch Hall
- Italy (5):
  - 1199.51.39002 Boehringer Ingelheim Investigational Site, Ancona
  - 1199.51.39001 Boehringer Ingelheim Investigational Site, Genova
  - 1199.51.39004 Boehringer Ingelheim Investigational Site, Macerata
  - 1199.51.39005 Boehringer Ingelheim Investigational Site, Reggio Emilia
  - 1199.51.39003 Boehringer Ingelheim Investigational Site, Udine
- Spain (6):
  - 1199.51.34007 Boehringer Ingelheim Investigational Site, A Coruña
  - 1199.51.34006 Boehringer Ingelheim Investigational Site, Alicante
  - 1199.51.34005 Boehringer Ingelheim Investigational Site, Barakaldo
  - 1199.51.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1199.51.34003 Boehringer Ingelheim Investigational Site, Madrid
  - 1199.51.34004 Boehringer Ingelheim Investigational Site, Madrid

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Maximum Tolerable Dose set (MTD): The first 12-18 patients randomised to the nintedanib treatment group, treated with nintedanib according to the dose escalation part of the study.
  The patient randomised to MTD analysis set were in Phase-1. The final data base lock date for this study was 23 JUL 2013.
Groups:
- Nintedanib 150 mg + mFolfox6: Patients receiving nintedanib 150 mg twice daily in a form of a soft gelatine capsule plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion).
- Nintedanib 200 mg + mFolfox6: Patients receiving nintedanib 200 mg twice daily in a form of a soft gelatine capsule plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion).
- Bevacizumab 5 mg + mFolfox6 (Phase II): Patients receiving bevacizumab 5 mg/kg every other week in a form of a bottles (injection concentrate solution) plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion).
Period: Overall Study
Arm/Group | Nintedanib 150 mg + mFolfox6 | Nintedanib 200 mg + mFolfox6 | Bevacizumab 5 mg + mFolfox6 (Phase II)
Started | 4 (All 4 patients were randomised to Maximum Tolerable Dose analysis set.) | 82 (11 patients were randomised to Maximum Tolerable Dose analysis set.) | 42 (Randomised)
Completed | 3 | 64 | 27
Not Completed | 1 | 18 | 15
Not completed — Adverse Event | 0 | 5 | 4
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Not treated | 1 | 0 | 1
Not completed — Other than above | 0 | 9 | 7

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) - The treated set includes all patients who were dispensed and were documented to have taken at least one dose of the trial drug.
Groups:
- Nintedanib + mFolfox6: Patients receiving nintedanib 150 mg or 200 mg twice daily in a form of a soft gelatine capsule plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion).
- Bevacizumab + mFolfox6: Patients receiving bevacizumab 5 mg/kg every other week in a form of a bottles (injection concentrate solution) plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion).
- Total: Total of all reporting groups
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6 | Total
Number analyzed (Participants) | 85 | 41 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.83) | 63.0 (9.36) | 62.8 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 21 | 60
  Male | 46 | 20 | 66

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 9 Months (PFS-9)
Description: PFS-9 is defined as the time from first treatment with the trial drug until either the onset of progressive disease or death. A patient is defined as progression-free for 9 months if their PFS was at least 270 days. Progression is assessed according to following mentioned RECIST criteria (version 1.0).
  1. 20% increase in the sum of the longest diameter of target lesions.
  2. The appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: First treatment administration to nine months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
percentage of Participants | 62.1 [50.2 to 73.9] | 70.2 [54.5 to 85.8]
Statistical Analysis 1: Comparison: Nintedanib + mFolfox6 vs Bevacizumab + mFolfox6; Test type: Superiority or Other; Kaplan-Meier; Difference = -8.1, 95% CI 2-sided [-27.8 to 11.5] — Difference in Kaplan-Meier Progression-free Survival Rates at 9 Months using Peto´s variance estimate

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from first treatment until death. Greenwood variance was used for the calculation of 95% confidence interval.
Time Frame: First treatment administration until end of treatment, up to 892 days
Population: Treated Set (TS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
months | 27.8 [24.5 to 30.8] | 33.4 [22.4 to NA] — Upper confidence limit for median cannot be estimated (i.e. the confidence limits does not extend beyond the last failure time).

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from first treatment with the trial drug until either the onset of progressive disease or death throughout the whole study. Progression is assessed according to RECIST criteria (version 1.0). In this endpoint, the Greenwood's variance estimate was used to calculate the Kaplan-Meier progression free survival median and its corresponding 95% confidence interval
Time Frame: First treatment administration until end of treatment, up to 892 days
Population: Treated Set (TS).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
months | 10.5 [9.4 to 12.4] | 15.4 [9.6 to 18.9]

4. Secondary Outcome: Confirmed Objective Response Rate
Description: Objective response rate is defined as a best response of either complete (CR) or partial response (PR) according to RECIST version 1.0. To be assigned a status of PR or CR, changes in tumour measurements had to be confirmed by repetition of the CT or MRI scan no less than 4 weeks after the criteria for response were first met. This confirmation was necessary to avoid overestimating the response rate observed. The 95% confidence interval represent the Clopper-Pearson exact confidence interval
Time Frame: First treatment administration until end of treatment, up to 892 days
Population: Treated Set (TS).
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
percentage of Participants | 63.5 [52.4 to 73.7] | 56.1 [39.7 to 71.5]

5. Secondary Outcome: Unconfirmed Objective Response Rate
Description: Objective response is defined as a best response of either complete (CR) or partial response (PR) according to RECIST version 1.0. To be assigned a status of PR or CR, changes in tumour measurements had to be confirmed by repetition of the CT or MRI scan no less than 4 weeks after the criteria for response were first met. This confirmation was necessary to avoid overestimating the response rate observed. The 95% Confidence interval represent the Clopper- Pearson exact confidence interval.
Time Frame: First treatment administration until end of treatment, up to 892 days
Population: Treated Set (TS).
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
percentage of Participants | 69.4 [58.5 to 79.0] | 73.2 [57.1 to 85.8]

6. Secondary Outcome: Resection Rate
Description: Surgical excision of the lesions is allowed if the previous assessment of tumoral response occurred after at least 6 cycles of treatment. Resection Rate includes resection rates R0, R1 and R2 before progressive disease.
  Peto's variance estimate was used.
Time Frame: First treatment administration until end of treatment, up to 892 days
Population: Treated Set (TS)
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
percentage of Participants | 19.5 [13.0 to 26.0] | 24.5 [16.6 to 32.4]
Statistical Analysis 1: Comparison: Nintedanib + mFolfox6 vs Bevacizumab + mFolfox6; Test type: Superiority or Other; Kaplan-Meier; Difference = -5.0, 95% CI 2-sided [-15.3 to 5.2] — confidence interval includes 0, meaning that the null hypothesis (no difference between the 2 groups) cannot be rejected (i.e. pvalue > 0.05). The pvalue was not computed. Difference in Kaplan-Meier Resection Rates using Peto´s variance estimate

7. Secondary Outcome: Tumor Shrinkage
Description: For each patient, the minimum percentage increase from baseline measurement (≤ 28 days before the beginning of the treatment) of the sum Longest diameter (LD) of target lesions was calculated based on the measurements of tumor size. The minimum percentage increase has been divided to four groups:
  1. <= - 30%
  2. > - 30% and < 0%
  3. >= 0% and < 20%
  4. >=20%
Time Frame: Baseline and day 85
Population: Treated Set (TS)
Measure: Number; unit: participants
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
participants
  <=-30% | 58 | 29
  > - 30% and < 0% | 19 | 7
  >= 0% and < 20% | 4 | 4
  >=20% | 2 | 0
  Non-evaluable | 2 | 1

8. Secondary Outcome: Incidence and Intensity of Adverse Events With Grading According CTCAE
Description: Incidence and intensity of Adverse Events with grading according to the Common Terminology Criteria for Adverse Events (CTCAE version 3.0).
Time Frame: From the first dose of study medication up to 28 days after the day of the last intake of study medication, up to 920 days
Population: Treated Set (TS)
Measure: Number; unit: participants
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
participants
  CTCAE Grade 1 | 1 | 0
  CTCAE Grade 2 | 9 | 2
  CTCAE Grade 3 | 62 | 29
  CTCAE Grade 4 | 11 | 7
  CTCAE Grade 5 | 2 | 3

9. Secondary Outcome: Percentage of Patients With Dose Limit Toxicity (DLTs) Incidence During the First Two Treatment Cycles (Phase I).
Description: Percentage of patients with DLTs,AE were observed in Gastrointestinal,Hepatobiliary & skin and subcutaneous tissue disorder.Drug related DLT was defined:1)Gastrointestinal toxicity(vomiting, nausea and diarrhoea)or hypertension of CTCAEgrade(G)3 despite optimal supportive care/intervention.2)Non-haematological toxicity of G≥3 except AE:alopecia,nail modifications,& isolated elevation of gamma glutamyl transpeptidase.3)G4 neutropenia for>7days(not associated with fever≥38.5°C).4)Neutropenia of G≥3 of any duration associated with fever≥38.5ºC.5)Platelets <25,000/μLorG3 thrombocytopenia associated with bleeding requiring transfusion.6)Inability to resume nintedanib dosing within14days of stopping due to treatment related toxicity.7)ALT and/or AST elevation of G≥3orG≥2 in conjunction with bilirubin G>1. 8)Inability to recover from increase ALT/AST in conjunction with increase of bilirubin toALT/AST toG≤1 &bilirubin to normal or baseline within14days after nintedanib treatment interruption
Time Frame: First two treatment cycles, up to 28 days
Population: MTD set: The first 12-18 patients randomised to the nintedanib treatment group, treated with nintedanib according to the dose escalation part of the study. The outputs (updated with cleaned and more complete data) that were used to decide on the MTD of nintedanib while the study was ongoing.
Measure: Number; unit: percentage of participants
Groups:
- Nintedanib 150 mg + mFolfox6 (Phase I): Patients receiving nintedanib 150 mg twice daily in a form of a soft gelatine capsule plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion)
- Nintedanib 200 mg + mFolfox6 (Phase I): Patients receiving nintedanib 200 mg twice daily in a form of a soft gelatine capsule plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion).
Arm/Group | Nintedanib 150 mg + mFolfox6 (Phase I) | Nintedanib 200 mg + mFolfox6 (Phase I)
Number analyzed (Participants) | 3 | 9
percentage of participants
  Diarrhoea | 0.0 | 11.1
  Hepatotoxicity | 0.0 | 11.1
  Rash maculo-papular | 33.3 | 0.0

10. Secondary Outcome: Maximum Tolerable Dose (MTD)
Description: Determination of Maximum Tolerable Dose based on DLT incidence.
Time Frame: First two treatment cycles, up to 28 days
Population: MTD Set
Measure: Number; unit: mg
Arm/Group | Nintedanib 150 mg + mFolfox6 (Phase I) | Nintedanib 200 mg + mFolfox6 (Phase I)
Number analyzed (Participants) | 3 | 9
mg | 200 | 200

11. Secondary Outcome: Area Under the Plasma Concentration Time-curve Over 12 Hours for Nintedanib in the Dosing Interval at Steady State and Normalized by the Dosing Unit Administered (AUCtau,ss,Norm) (Phase I)
Description: Area under the plasma concentration time-curve over 12 hours for Nintedanib in the dosing interval at steady state and normalized by the dosing unit administered (AUCtau,ss,norm) (Phase I)
Time Frame: -0:05h before drug administration and 1h, 2h, 2.5h, 3h, 4h, 6h, 8h and 10h after drug administration.
Population: Treated Set (TS).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Nintedanib 150 mg + mFolfox6 (Phase I) | Nintedanib 200 mg + mFolfox6 (Phase I)
Number analyzed (Participants) | 3 | 4
ng*h/mL/mg | 1.46 (273) | 1.53 (30.1)

12. Secondary Outcome: Maximum Plasma Concentration for Nintedanib at Steady State and Normalized by the Dosing Unit Administered (Cmax,ss,Norm) (Phase I)
Description: Maximum plasma concentration for Nintedanib at steady state and normalized by the dosing unit administered (Cmax,ss,norm) (Phase I)
Time Frame: -0:05h before drug administration and 1h, 2h, 2.5h, 3h, 4h, 6h, 8h, and 10h after drug administration.
Population: Treated Set (TS).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Nintedanib 150 mg + mFolfox6 (Phase I) | Nintedanib 200 mg + mFolfox6 (Phase I)
Number analyzed (Participants) | 3 | 5
ng/mL/mg | 0.294 (319) | 0.278 (34.0)

13. Secondary Outcome: Quality of Life Evaluation by a Standardised Questionnaires of EORTC: EORTC-QLQ-C30 for the Change From Baseline at 9 Months of Global Health Status Scores.
Description: Quality of life evaluation by a standardised questionnaires of European Organisation for Research and Treatment of Cancer (EORTC): EORTC-QLQ-C30 for the change from baseline at 9 months for Global health status scores.
  Raw scores are transformed to scales of 0-100. A higher score is associated with a better quality of life for Global health status scores
Time Frame: Baseline and 9 months.
Population: Treated Set (TS). Number of analysed patients are the total number of patients who were analysed for the change from baseline at 9 months for Global health status scores
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 24 | 11
units on scale | -1.7 (19.3) | -9.8 (13.9)

14. Secondary Outcome: Quality of Life Evaluation by a Standardised Questionnaires of EORTC: EORTC-QLQ-CR38 for the Change From Baseline at 9 Months.
Description: Quality of life evaluation by a standardised questionnaires of European Organisation for Research and Treatment of Cancer (EORTC): EORTC-QLQ-CR38 for the change from baseline at 9 months for functional scales, Symptom scales Chemotherapy side effects .
  The EORTC-QLQ-CR38 was composed of functioning scales (body image, future perspective, sexual enjoyment, sexual functioning) and symptom scales (chemotherapy side effects, defecation problems, symptoms of the gastrointestinal tract, micturition problems,female sexual problems, male sexual problems, stoma related problems, and weight loss).
  Raw scores are transformed to scales of 0-100. A higher score is associated with a better quality of life for functional scales and a worse quality of life for symptom scales.
Time Frame: Baseline and 9 months.
Population: Treated Set (TS)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 83 | 41
units on scale
  Body image (N=24, 11) | -3.2 (25.3) | -3.5 (19.0)
  Future perspective (N=25, 11) | 22.7 (35.6) | 6.1 (36.0)
  Sexual enjoyment (N=2, 3) | -33.3 (47.1) | -11.1 (19.2)
  Sexual functioning (N=15, 7) | -11.1 (17.4) | 2.4 (11.5)
  Chemotherapy side effects (N=25, 11) | 20.0 (30.9) | 13.1 (13.9)
  Defaecation problems (N=17, 8) | -5.4 (20.8) | 2.0 (7.7)
  Female sexual problems (N=0, 0) | NA (NA) — There was no patient reported for this scale | NA (NA) — There was no patient reported for this scale
  Male sexual problems (N=5, 4) | 6.7 (49.4) | 4.2 (16.0)
  Micturition problems (N=25,11) | -5.8 (21.1) | -7.1 (18.1)
  Stoma-related problems (N=4, 2) | -4.8 (10.3) | 2.4 (3.4)
  Symptoms area of gastro-intestinal tract (N=25,11) | -3.0 (13.3) | 3.4 (15.0)
  Weight loss (N=25,11) | -21.3 (31.7) | -12.1 (47.8)

15. Secondary Outcome: Number of Participants for Quality of Life Evaluation by a Standardised Questionnaires of EORTC: EORTC-QLQ-CR38 for the First Use of Stoma Bag.
Description: Number of participants for Quality of life evaluation by a standardised questionnaires of European Organisation for Research and Treatment of Cancer (EORTC): EORTC-QLQ-CR38 for the first use of stoma bag.
Time Frame: from baseline until end of treatment, up to 892 days
Population: Treated Set (TS).
Measure: Number; unit: participants
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Number analyzed (Participants) | 85 | 41
participants
  Baseline | 10 | 4
  Week 6 | 3 | 0
  Week 12 | 1 | 0
  Week 24 | 1 | 0
  Week 30 | 1 | 0
  Week 54 | 1 | 0
  No use of stoma bag | 68 | 37

16. Secondary Outcome: Exploratory Biomarker and Pharmacogenetic Analysis for VEGF
Description: Exploratory biomarker and pharmacogenetic analysis for Vascular endothelial growth factor (VEGF).
  Note: This endpoint was not statistically analysed in this study.
Time Frame: Day 1, Day 29, Day 57, Day 85 and Day 127
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first dose of study medication up to 28 days after the day of the last intake of study medication, up to 920 days
Groups:
- Nintedanib + mFolfox6: Patients receiving nintedanib 150 mg or 200 mg twice daily plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion).
- Bevacizumab + mFolfox6: Patients receiving bevacizumab 5 mg/kg every other week plus mFolfox6: oxaliplatin 85 mg/m², l-leucovorin 200 mg/m² or d, l-leucovorin 400 mg/m², 5-fluorouracil 400 mg/m² (bolus) and 2400 mg/m² (infusion)
Arm/Group | Nintedanib + mFolfox6 | Bevacizumab + mFolfox6
Serious Adverse Events (participants affected / at risk) | 31/85 | 22/41
Other Adverse Events (participants affected / at risk) | 84/85 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib + mFolfox6 (N=85) | Bevacizumab + mFolfox6 (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Intestinal perforation (Gastrointestinal disorders) | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Condition aggravated (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Prosthesis implantation (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib + mFolfox6 (N=85) | Bevacizumab + mFolfox6 (N=41)
Anaemia (Blood and lymphatic system disorders) | 11 | 2
Neutropenia (Blood and lymphatic system disorders) | 38 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 3
Vertigo (Ear and labyrinth disorders) | 5 | 0
Abdominal pain (Gastrointestinal disorders) | 18 | 8
Abdominal pain upper (Gastrointestinal disorders) | 13 | 7
Constipation (Gastrointestinal disorders) | 16 | 19
Diarrhoea (Gastrointestinal disorders) | 63 | 25
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Flatulence (Gastrointestinal disorders) | 4 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 60 | 24
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 4
Stomatitis (Gastrointestinal disorders) | 13 | 6
Toothache (Gastrointestinal disorders) | 0 | 5
Vomiting (Gastrointestinal disorders) | 37 | 12
Asthenia (General disorders) | 47 | 25
Chest pain (General disorders) | 5 | 1
Chills (General disorders) | 2 | 3
Fatigue (General disorders) | 26 | 11
Mucosal inflammation (General disorders) | 18 | 16
Oedema peripheral (General disorders) | 4 | 4
Pain (General disorders) | 6 | 1
Pyrexia (General disorders) | 14 | 10
Drug hypersensitivity (Immune system disorders) | 6 | 4
Nasopharyngitis (Infections and infestations) | 8 | 5
Urinary tract infection (Infections and infestations) | 6 | 2
Alanine aminotransferase increased (Investigations) | 5 | 1
Gamma-glutamyltransferase increased (Investigations) | 5 | 2
Weight decreased (Investigations) | 8 | 4
Decreased appetite (Metabolism and nutrition disorders) | 26 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 6 | 6
Dysaesthesia (Nervous system disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 16 | 5
Headache (Nervous system disorders) | 6 | 5
Neuropathy peripheral (Nervous system disorders) | 16 | 7
Neurotoxicity (Nervous system disorders) | 19 | 13
Paraesthesia (Nervous system disorders) | 31 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 3
Polyneuropathy (Nervous system disorders) | 8 | 3
Depression (Psychiatric disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 5 | 8
Haematuria (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 5
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 | 9
Rash (Skin and subcutaneous tissue disorders) | 6 | 1
Hypertension (Vascular disorders) | 15 | 11
Hypertensive crisis (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights